CLINICAL TRIAL: NCT02753439
Title: Extraction of Impacted 3rd Molars, Can Bone Support of the Second Molar be Promoted by a Bio-Oss Graft?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Baruchpmc.CTIL
Record Dates: First submitted 2016-03-20; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3rd molar (Experimental): Drug: Geistlich Bio Oss
  Interventions: Drug: Geistlich Bio Oss

INTERVENTIONS:
Drug: Geistlich Bio Oss — Extraction of Impacted 3rd Molars,
  Other Names: Bone Support

SUMMARY:
A prospective study examining bilateral 3rd molar extraction, by a split mouth protocol the investigators augment unilaterally and compare periodontal parameters in between.

DETAILED DESCRIPTION:
40 patients will undergo bilateral 3rd molar extractions, in each patient one side would be augmented by a "Bio-Oss" xenograft.

Post operative, periodontal parameters such as pocket depth and mobility will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral impacted 3rd molars.
* Healthy individuals

Exclusion Criteria:

* Smokers
* Alcohol abusers
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Mobility (Scale 0,1,2,3), change is being assessed. | Pre opp (base line), 1 month post opp, 3 months post opp, 6 months post opp
  Mobility will be assessed in the intervals mentioned above, and compared over time.
Pocket Depth (mm), change is being assessed. | Pre opp (base line), 1 month post opp, 3 months post opp, 6 months post opp
  Pocket depth will be assessed in the intervals mentioned above, and compared over time.

IPD SHARING:
Plan to Share IPD: No